CLINICAL TRIAL: NCT00117481
Title: A Phase 2, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate DR-2001 for the Management of Moderate to Severe Endometriosis-Related Nonmenstrual Pelvic Pain
Brief Title: Evaluation of DR-2001 for the Management of Endometriosis-Related Pelvic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-DZL-201
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Endometriosis
Keywords: endometriosis; pelvic pain; hormonal treatment
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: DR-2001a
- 2 (Experimental)
  Interventions: Drug: DR-2001b
- 3 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DR-2001a — DR-2001a administered vaginally each month
  Arms: 1
Drug: DR-2001b — DR-2001b administered vaginally each month
  Arms: 2
Other: Placebo — Placebo administered vaginally each month
  Arms: 3

SUMMARY:
This is a 3-arm, multicenter, double-blind, randomized, placebo-controlled study to evaluate the efficacy of DR-2001 in endometriosis-related symptoms, primarily nonmenstrual pelvic pain, over a 12-week treatment period.

DETAILED DESCRIPTION:
This multicenter, double-blind, randomized, placebo-controlled study is designed to evaluate the ability of DR-2001 to produce beneficial changes in endometriosis-related symptoms, primarily nonmenstrual pelvic pain, over a 12-week treatment period. The overall study duration for each patient will be about 20 weeks.

Patients who meet all study entrance criteria will be randomly assigned to one of three treatment groups.

The change in endometriosis-related clinical symptoms will be assessed in two ways: through a combined physician/patient assessment and also with a patient self-assessment. Patients will undergo a gynecologic exam at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Surgically sterilized (patient or partner), willing to use condoms throughout the study, or otherwise not at risk for pregnancy
* Diagnosis of endometriosis within the last 5 years
* Moderate or severe nonmenstrual pelvic pain
* Premenopausal
* Not pregnant or breastfeeding
* Regular (24-35 day) menstrual cycles for at least 2 months

Exclusion Criteria:

* Undiagnosed abnormal genital bleeding
* Any contraindication to the use of hormonal therapy
* Prior surgery for endometriosis
* GnRH analog therapy within 5 months
* Use of estrogens and/or progestins within 2 months
* Pain symptoms unrelated to endometriosis
* Any contraindication to the use of vaginal delivery systems

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Mean change in nonmenstrual pelvic pain at end of treatment | Baseline to Week 12/Early Withdrawal Visit

SECONDARY OUTCOMES:
Mean change in nonmenstrual pelvic pain and endometriosis-related symptoms | Weeks 4, 8 and 12
Safety and tolerability of DR-2001 | Throughout study period

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (41):
- United States (41):
  - Duramed Investigational Site, Enterprise, Alabama
  - Duramed Investigational Site, Montgomery, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Little Rock, Arkansas
  - Duramed Investigational Site, La Jolla, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Vista, California
  - Duramed Investigational Site, Colorado Springs, Colorado
  - Duramed Investigational Site, Clearwater, Florida
  - Duramed Investigational Site, Hudson, Florida
  - Duramed Investigational Site, Spring Hill, Florida
  - Duramed Investigational Site, Tampa, Florida
  - Duramed Investigational Site, West Palm Beach, Florida
  - Duramed Investigational Site, Decatur, Georgia
  - Duramed Investigational Site, Idaho Falls, Idaho
  - Duramed Investigational Site, La Grange Park, Illinois
  - Duramed Investigational Site, Maywood, Illinois
  - Duramed Investigational Site, Oak Brook, Illinois
  - Duramed Investigational Site, Louisville, Kentucky
  - Duramed Investigational Site, Ann Arbor, Michigan
  - Duramed Investigational Site, Reno, Nevada
  - Duramed Investigational Site, Princeton, New Jersey
  - Duramed Investigational Site, Port Jefferson, New York
  - Duramed Investigational Site, Chapel Hill, North Carolina
  - Duramed Investigational Site, Morganton, North Carolina
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Dayton, Ohio
  - Duramed Investigational Site, Oklahoma City, Oklahoma
  - Duramed Investigational Site, Jenkintown, Pennsylvania
  - Duramed Investigational Site, Florence, South Carolina
  - Duramed Investigational Site, Jackson, Tennessee
  - Duramed Investigational Site, Memphis, Tennessee
  - Duramed Investigational Site, Austin, Texas
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Pleasant Grove, Utah
  - Duramed Investigational Site, Sandy City, Utah
  - Duramed Investigational Site, Norfolk, Virginia
  - Duramed Investigational Site, Virginia Beach, Virginia